CLINICAL TRIAL: NCT03212937
Title: A Phase I Investigator Sponsored Trial of Selinexor (KPT-330), a Selective Inhibitor of Nuclear Export / SINE™ Compound and Ifosfamide, Carboplatin, Etoposide (ICE) in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: Phase I Trial of Selinexor (KPT-330) and Ifosfamide, Carboplatin, Etoposide (ICE) in Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Karyopharm001
Record Dates: First submitted 2017-06-28; First posted 2017-07-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — selinexor; ICE protocol 5; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor and ICE Chemotherapy (Experimental)
  Interventions: Drug: Selinexor; Drug: ICE Chemotherapy

INTERVENTIONS:
Drug: Selinexor — Oral KPT-330 is administered on Day 3, 5, and 7 of each 21-day cycle. Starting dose is 40mg will be adjusted according to toxicity
Drug: ICE Chemotherapy — IV Ifosfamide 5g/m^2 on Day 2 (inpatient) or D1 (outpatient) of each 21-day cycle
  IV Carboplatin AUC 5 on Day 2 (inpatient) or D1-3 (outpatient) of each 21-day cycle
  IV Etoposide 100 mg/m^2 on Days 1-3 of each 21-day cycle
  Other Names: Ifosfamide, Carboplatin, Etoposide

SUMMARY:
This is a single center, open-label, phase I trial with a standard 3+3 dose escalation schema to identify the maximum tolerated dose (MTD) of selinexor when combined with ICE. Once MTD is determined, there will be an expansion phase and tumor biopsies and peripheral blood will be taken pre and post selinexor to examine the study's biologic objectives.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary:

• To determine the maximum tolerated dose (MTD) of selinexor when given in combination with a standard dose regimen of ifosfamide, carboplatin and etoposide (ICE) in patients with relapsed or refractory PTCL

Secondary:

* To assess the response rates (complete and partial), progression-free survival (PFS) and overall survival (OS) in patients with relapsed or refractory PTCL
* To estimate the feasibility of stem cell collection after selinexor and ICE

Laboratory objectives:

• Paired tumor specimens pre and post selinexor will be examined ex vivo for

* Response to chemotherapy agents such as doxorubicin and etoposide
* Nuclear localization of tumor suppressor proteins (p53, p73, FOXO), drug targets (topoisomerase II) and mRNA targets

STUDY DESIGN:

This is a single center, open-label, phase I trial with a standard 3+3 dose escalation schema to identify the maximum tolerated dose (MTD) of selinexor when combined with ICE. Once MTD is determined, there will be an expansion phase and tumor biopsies and peripheral blood will be taken pre and post selinexor to examine the study's biologic objectives.

Dose escalation:

* If 0/3 dose-limiting toxicity (DLT) is observed, dose escalation will continue to the next higher dose level.
* If 1/3 DLT is observed, then 3 additional patients will be enrolled in the same dose level; if no DLT is observed from the additional 3 patients, then dose escalation will continue to the next higher dose level. If any DLT is observed from the additional 3 patients, then the previous lower dose will be chosen as the MTD.
* If ≥ 2/3 DLTs are observed, then the previous lower dose level will be chosen as the MTD and the dose finding procedure will be terminated.

PATIENTS:

Subjects will be enrolled at the National Cancer Centre Singapore (NCCS).

Key eligibility criteria include the following:

* Pathologically confirmed aggressive T-cell lymphomas including the following histologies: PTCL-NOS, AITL, ALCL (independent of ALK status), NK/T-cell lymphoma
* Treatment with at least two cycles of one prior regimen administered with curative intent
* Adequate end-organ and bone marrow function
* Absence of known or suspected CNS involvement
* Absence of active viral hepatitis or uncontrolled HIV

STUDY DURATION:

Based on prior and existing patient volumes and accrual to clinical trials, we expect to enroll 1-2 patients per month. We expect to complete study accrual within 2 years.

TOTAL SAMPLE SIZE:

The MTD will be identified using a standard 3+3. A maximum of 18 patients will be required for this phase I study. An additional 5 patients will be treated at the recommended phase II dose to assess safety and to examine the study's biologic objectives.

DOSING REGIMEN:

Dose escalation schedule for selinexor:

Dose level -1: 20mg

Dose level 1: 40mg

Dose level 2: 60mg

Dose level 3: 80mg

Selinexor will be administered on days 3, 5 and 7 of each chemotherapy cycle and ICE will be administered from day 1. In the expansion phase of the study, selinexor is administered on days -5 and -3 prior to cycle 1 of chemotherapy.

All subjects will receive

(I) Standard dose ICE on a 21-day cycle.

* IV Etoposide 100mg/m^2 on D1-3
* IV Carboplatin AUC 5 on D2 (inpatient) or D1 (outpatient)
* IV Ifosfamide 5g/m^2 on D2 (inpatient) or D1-3 (outpatient)

(II) Dexamethasone

* 20mg QD D3-7
* 20mg QD D-5 and D-3 (for patients in the expansion phase)

Patients will receive 2-6 cycles of selinexor and ICE. If determined eligible by their treating physician, patients who demonstrate response will undergo autologous stem cell transplantation anytime following the second cycle of selinexor and ICE. Transplant ineligible patients will complete up to 6 cycles of selinexor and ICE, and those with responses or stable disease are eligible for maintenance selinexor at the discretion of the treating physician. Maintenance selinexor will be administered weekly at the dose of 60mg. Dexamethasone 4-12mg should also be given on the selinexor dosing days.

ASSESSMENT:

CT Neck to pelvis or FDG-PET/CT skull base to mid-thigh to be performed repeated after every 2 cycles on days 17 +/- 3 days except after cycle 2 where FDG-PET/CT will be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed T or NK/T-cell lymphomas including the following histologies:

  * Peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS)
  * Angioimmunoblastic T-cell lymphomas (AITL)
  * Anaplastic large cell lymphoma (ALCL)
  * Natural-killer/T-cell lymphoma (NKTL)
* Patients must have received at least two cycles of one prior regimen administered with curative intent and one of the following:

  * failed to have achieve at least a partial response after 2 or more cycles
  * failed to achieve a complete response after 6 or more cycles
  * progressed after an initial response
  * For patients who have CD30+ anaplastic large cell lymphoma, they must have failed or are ineligible or intolerant of brentuximab vedotin
* Patients must be age >18 years.
* Patients must have at least one site of measurable disease, 1.5 cm in diameter or greater.
* Patients must have ECOG performance status of 0-2
* Patients must have laboratory test results within these ranges:

  * Absolute neutrophil count ≥1500/mm³
  * Platelet count ≥75,000/mm³
  * Creatinine clearance ≥40ml/min
  * Total bilirubin ≤1.5x ULN. Higher levels are acceptable if these can be attributed to active haemolysis or ineffective erythropoiesis.
  * AST (SGOT) and ALT (SGPT) ≤2x ULN
* Women of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test prior to KPT-330 treatment. Male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential.

  * Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal.
  * For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.

As the effects of selinexor on the developing human fetus at the recommended therapeutic dose are unknown, women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with selinexor. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women that are pregnant or breastfeeding are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

* Patients must be able to understand and willing to sign a written informed consent document.
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patients must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

Exclusion Criteria:

* Patients who have had prior malignancies (other than T and NK/T-cell lymphomas) for ≤5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Patients who have had other anti-cancer therapy, including radiation or experimental drug or therapy, within 28 days of enrollment.
* Patients with known HIV, active hepatitis B, active hepatitis C.
* Patients with known central nervous system involvement by lymphoma.
* Patients with known or suspected hypersensitivity to selinexor.

Inclusion of Women and Minorities:

Men and women of all ethnic groups are eligible for this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related dose limiting toxicity as assessed by NCI CTCAE v4.0 | The first 3 weeks of treatment

SECONDARY OUTCOMES:
Overall response rate | From the start of treatment to the best overall response of Complete or Partial Response is achieved, up to 2 years
  Responses will be assessed using the revised International Workshop Criteria
Progression-free survival | From the start of the treatment to the date of documentation of either disease progression or death, up to 2 years
Overall survival | From the start of treatment to the date of death from any cause, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany PL Tang, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No